CLINICAL TRIAL: NCT06780878
Title: Comparison of Progressive Muscle Relaxation and Stretching Exercises Mediated by Stress in Diabetic Population
Brief Title: Comparison of Progressive Muscle Relaxation and Stretching Exercises in Diabetic Population
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Rana Ghunwa Tanveer
Record Dates: First submitted 2025-01-13; First posted 2025-01-17 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Diabetes Mellitus Type 2
Keywords: perceived stress; progressive muscle relaxation; stretching exercises; heart rate variability; cortisol levels; galvanic skin response
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Muscle Stretching Exercises; Control Groups

STUDY DESIGN:
Intervention Model Description: The study consists of 2 active comparators and 1 control group.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Progressive muscle relaxation technique (Experimental): This group will consist of 12 female participants of age 35-65 years with Diabetes Mellitus type 2. This group will be given PMR, 10 minutes per session, 3 sessions per week for 2 weeks. Blood pressure (BP,) Blood sugar random (BSR), Oxygen saturation (SPO2), Heart rate (HR), Heart rate variability (HRV), Galvanic skin response (GSR), and Cortisol levels (CL) will be measured before and after every session. Perceived Stress Scale will be used to assess participants' stress levels at baseline and then after 2 weeks.
  Interventions: Other: Progressive muscle relaxation technique
- Stretching exercises (Experimental): This group will consist of 12 female participants of age 35-65 years with Diabetes Mellitus type 2. Participants will be given stretching exercises, 10 minutes per session, 3 sessions per week for 2 weeks. Blood pressure (BP,) Blood sugar random (BSR), Oxygen saturation (SPO2), Heart rate (HR), Heart rate variability (HRV), Galvanic skin response (GSR), and Cortisol levels (CL) will be measured before and after every session. Perceived Stress Scale will be used to assess participants' stress levels at baseline and then after 2 weeks.
  Interventions: Other: Stretching exercises
- Control group (Other): This group will consist of 12 participants who will not be given any physical therapy interventions. Same measurements will be taken at same intervals as the experimental groups.
  Interventions: Other: Control Group

INTERVENTIONS:
Other: Progressive muscle relaxation technique — PMR focuses on the relationship between muscle tension and relaxation. By deliberately tensing a muscle group for a few seconds and then releasing the tension, individuals become more aware of the sensation of relaxation.
  Group A Participants will receive PMR for 10 minutes each session, 3 sessions per week for 2 weeks and outcome measures will be recorded pre and post for each session.
  Arms: Progressive muscle relaxation technique
Other: Stretching exercises — Stretching exercises are physical activities designed to improve the flexibility of muscles and joints. These exercises involve elongating specific muscle groups to enhance their elasticity and improve the range of motion around a joint.
  Participants will be given 15 second stretches for each large muscle group, 3 sessions per week, for 2 weeks. Outcome measures will be assessed pre and post intervention.
  Arms: Stretching exercises
Other: Control Group — This group will consist of 12 participants who will not be given any physical therapy interventions. Same measurements will be taken at same intervals as the experimental groups.
  Arms: Control group

SUMMARY:
The goal of this clinical trial is to compare the effects of Progressive muscle relaxation and stretching exercises mediated by stress on heart rate variability, cortisol level, galvanic skin response and perceived stress scale. The main questions it aims to answer are, Will there be a significant difference between the effects of Progressive muscle relaxation and stretching exercises in the diabetic population? Can stress mediate the effects of Progressive muscle relaxation and stretching exercises in the diabetic population?

Researchers will compare the effects of Progressive muscle relaxation and stretching exercises mediated by stress on heart rate variability, cortisol level, galvanic skin response and perceived stress scale.

Participants will:

Be given session of Progressive muscle relaxation or stretching exercises or no physical therapy treatment 3 sessions per week for 2 weeks and visit the clinic once every 3 days for 2 weeks for intervention. Measurements will be taken before and after every session. Perceived Stress will be assessed at the start of the intervention at baseline and then after 2 weeks.

DETAILED DESCRIPTION:
The subject of this research is individuals with type 2 diabetes who also experience depression. Progressive muscle relaxation (PMR) has the potential to reduce blood sugar levels in type 2 diabetes patients. This reduction is linked to the stress, both physical and psychological, experienced by the patients.

When stressors are assessed, muscle tension is created, which signals the brain and creates a feedback. PMR works to interrupt this loop by stimulating the parasympathetic nervous system and influencing the hypothalamus through focused concentration, promoting a positive mindset and reducing stress on the hypothalamus. Stretching can also be easily integrated into a diabetic's daily routine promoting both physical and mental wellbeing.

Most studies focus on PMR or stretching exercises separately in managing stress, but comparing these two interventions in terms of stress reduction and physical outcomes in diabetics is limited.

Understanding which intervention provides better stress relief could lead to more targeted recommendations in diabetic care.

ELIGIBILITY:
Inclusion Criteria:

* Age 35-65 years
* Females
* Uncontrolled Diabetes Mellitus
* Sedentary Lifestyle
* Has never undergone progressive muscular relaxation before.

Exclusion Criteria:

* Unstable Angina
* Cardiac arrhythmia
* Postural deformities
* Left ventricular ejection fraction < 45%

Ages: 35 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Females are eligible to participate in the study.
Enrollment: 36 (Actual)
Dates: Start 2025-02-01 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Heart rate variability | 24 hours
  It is a valuable tool in various fields, including health, fitness, and psychology for assessing the body's physiological responses. HRV is linked to emotional regulation and mental health, lower HRV is often associated with anxiety, depression, and other mental health conditions. In therapeutic settings, biofeedback using HRV can help individuals learn to manage stress and improve emotional resilience. HRV has been validated as a tool to measure autonomic nervous system activity, particularly the balance between sympathetic(stress) and parasympathetic (recovery) responses it is widely used in stress and fatigue research. HRV shows good test-retest reliability when measured under consistent conditions, such as in the same environment at the same time, of the day, and in the same position.
Cortisol levels | 24 hours
  Cortisol is a hormone released in response to stress, typically measured through saliva or blood samples. CL is used to monitor how well a patient is responding to treatment for conditions like adrenal disorders depression, or stress related illness. It can be measured through saliva, blood, urine, and hair being a common non-invasive method. Cortisol is widely regarded as a valid indicator of physiological stress. Cortisol is sensitive to external factors including stressors like physical exertion or even the experience of being tested. The reliability of cortisol as a measure of stress or health depends heavily on stress control.
Galvanic skin response | 24 hours
  GSR also known as electro-dermal activity, is a physiological measure of skin conductance that reflects changes in sweat gland activity. GSR measures the skin's ability to conduct electricity. When a person experiences emotional arousal, the (SNS triggers sweat glands, particularly on the palms and soles to become more active, this increases the skin's electrical conductance which the GSR sensor can detect. GSR is generally considered valid in measuring arousal or emotional intensity It is a good indicator of stress, anxiety, or excitement because these emotions typically involve a heightened autonomic nervous system.
Perceived stress | 2 weeks
  Perceived stress scale is a widely used psychological instrument designed to assess the perception of stress. It helps to measure the degree to which situations in one's life are appraised as stressful. It evaluates the subjective experience of stress. Which can vary significantly between individuals. Studies have confirmed that the PSS effectively measures perceived stress, a psychological state characterized by feelings of unpredictability and uncontrollability. The Perceived Stress Scale (PSS) scoring involves summing the responses to 10 questions, with higher scores indicating higher perceived stress levels. The scale uses a 5-point Likert scale, where 0 represents "never" and 4 represents "very often". Some questions are reverse-scored to account for coping mechanisms. Scores can range from 0 to 40, with ranges like 0-13 (low), 14-26 (moderate), and 27-40 (high) used for general interpretation

CONTACTS AND LOCATIONS:
Overall Officials: Maria Naeem, DPT, MS-CPPT, Principal Investigator — Riphah International University
Locations (1):
- Pakistan Railway General Hospital, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No